CLINICAL TRIAL: NCT00075075
Title: Pilot Study of the Evaluation of Infliximab in the Treatment of Non-Infectious Scleritis
Brief Title: Infliximab to Treat Non-Infectious Scleritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040065; 04-EI-0065
Record Dates: First submitted 2003-12-31; First posted 2004-01-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-06

CONDITIONS: Scleritis
Keywords: Infliximab; Scleritis; Intraocular Inflammatory Disease; Corticosteroids; Immunosuppressives
MeSH Terms: conditions — Scleritis | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
This small, preliminary study will examine whether multiple infusions of infliximab (Remicade® (Registered Trademark)) can control inflammation in patients with active scleritis. The sclera is the tough white outer coat enclosing the eyeball. Infliximab is a combination of part human and part mouse proteins that block a natural body protein called tumor necrosis factor (TNF). TNF appears to be involved in scleritis, and stopping its action may help reduce the inflammation in the disease. The drug has been approved by the Food and Drug Administration for treating Crohn's disease and rheumatoid arthritis.

Patients 18 years of age or older with active non-infectious scleritis may be eligible for this study. Participants will undergo the following tests and procedures:

* Medical history and physical examination.
* Eye examination, including a vision test and examination of the retina (back part of the eye) and of the sclera and its blood vessels.
* Questionnaire about vision and daily activities.
* Tuberculin skin test.
* Pregnancy test: Women who can have children are tested for pregnancy at study weeks 0, 14, 30, 38, and 46.
* Infliximab treatment: Infliximab is infused over a 2-hour period through a needle in a vein, usually in the arm. The patient's vital signs are checked before the patient begins each infusion starts and again before leaving the clinic. After the first two infusions, if the disease remains quiet, other scleritis medications will be attempted to be reduced to half the original dose over 8 to 12 weeks and possibly to nothing if the patient continues to do well. Patients receive a maximum of 9 infusions over a 30-week period.
* Blood draws: About 4 tablespoons of blood are drawn at each visit to test for the number and types of cells in the blood and to check for signs of inflammation and side effects of the study medicine.

Patients are seen in the NEI clinic for infusions and to check the response to therapy. This includes 13 clinic visits over 46 weeks, as follows: every 2 weeks for the first 2 weeks, every 4 weeks thereafter for a total of 30 weeks for infusions, and then every 4 weeks for 16 additional weeks.

Patients may stop therapy if their scleritis is not controlled 10 weeks into the study period; if they develop a flare of inflammation after initial control of the active scleritis; if their vision loss is too large; or if their medications increase or other medicines are added to control the scleritis. Patients whose vision decreases minimally, stays the same, or improves may remain in the study.

DETAILED DESCRIPTION:
We propose to investigate the possible efficacy of multiple infliximab infusions to control the inflammation in participants presenting with active scleritis. This will be performed using an open-label pilot study. Subjects will receive 5mg/kg intravenous infusions of infliximab at 0, 2, 6 and 10 weeks. After these initial infusions, participants may contine to receive 5 mg/kg dose infusions or may receive 8 mg/kg dose infusions depending on the treamtent response. Treatment response is defined as a decrease in inflammation by at least 2 steps on the scale of grades 0-4 , or a decrease to 0 assessed at week 14. A combination of thse two dose infusions (5 mg/kg or 8 mg/kg) will be given for the remainder of the study according to set schedules. The primary outcome will be the ability to control active scleritis defined as at least a 2-step decrease in sleral inflammation,scleritis within 14 weeks of initiating infliximab therapy. Secondary outcomes will be the amount of reduction in concomitant immunosuppressive medication (measured using the grading scale in Section 4.5.2), changes in pain, redness (measured using a visual analogue scale), photophobia, changes in visual acuity (changes of 10 letters from baseline in best-corrected visual acuity will be considered clinically significant), the typical time between flares, and numbers of flares and times between flares while in the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to enroll in this study, a prospective participant must satisfy the following inclusion criteria:

1. Participant is 18 years of age or older.
2. Participant has active non-infectious scleritis, diagnosed by a persistent congestion of deep episcleral vessels following a drop of 10% phenylephrine, without active intraocular inflammation.
3. Participant has normal renal or liver function.
4. Participant agrees to use acceptable birth control methods throughout the course of the study and for 6 months after completion of treatment.
5. Participant has no evidence of tuberculosis as documented by tuberculin skin test performed prior to enrollment (chest x-ray, if medically indicated).
6. Participant is able to understand and sign a consent form before entering the study.
7. Participant has been treated with prednisone or other immunomodulatory medications but present with active disease at the time of enrollment.

EXCLUSION CRITERIA:

To be eligible to enroll in this study, a prospective participant must not satisfy any of the following exclusion criteria:

1. Participant with a known underlying systemic disease with evidence of serious or potentially lethal uncontrolled active disease in one or more extraocular organ systems for which a defined effective medical regimen is indicated.
2. Participant with a corneal melting, necrotizing keratitis, or impending vision loss.
3. Participant with scleritis of infectious etiology.
4. Participant receiving any other investigational therapy or another anti-TNF agent that would interfere with the ability to evaluate the safety or efficacy of infliximab.
5. Participant has significant active infection requiring hospitalization.
6. Participant with multiple sclerosis.
7. Participant has severe (class 3/4) congestive heart failure.
8. Participant has a history of cancer within the past 5 years other than basal or squamous cell carcinoma.
9. Participant is pregnant or lactating as it is unknown whether infliximab is excreted in human milk or absorbed systemically after ingestion.
10. Evidence of liver disease (any etiology).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2003-12-23; Study Completion 2007-09-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nguyen QD, Foster CS. Scleral patch graft in the management of necrotizing scleritis. Int Ophthalmol Clin. 1999 Winter;39(1):109-31. doi: 10.1097/00004397-199903910-00011. PMID 10083910